CLINICAL TRIAL: NCT02086344
Title: The Effect in Term of Ovarian Reserve Modification of Adding Prophylactic Bilateral Salpingectomy (PBS) to TLH for Preventing Ovarian Cancer
Brief Title: Ovarian Reserve Modification After Lps Hysterectomy With Bilateral Salpingectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full Professor Obstetric Gynecology, University Magna Graecia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PBS_hysterectomy
Record Dates: First submitted 2014-03-09; First posted 2014-03-13 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Uterine Fibroids; Adenomyosis; Pelvic Pain; Pelvic Prolapse
Keywords: Total Laparoscopic Hysterectomy; TLH; Ovarian reserve; Prophylactic bilateral salpingectomy; Ovarian cancer prevention; Ovarian cancer; Fallopian Tubes
MeSH Terms: conditions — Leiomyoma; Adenomyosis; Pelvic Pain; Ovarian Neoplasms | interventions — Salpingectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TLH_plus_PBS (Experimental): TLH plus PBS
  Interventions: Procedure: PBS
- TLH _adnexal preservation (Active Comparator): Standard TLH without PBS
  Interventions: Procedure: TLH _adnexal preservation

INTERVENTIONS:
Procedure: PBS — TLH plus PBS
  Other Names: Bilateral Salpingectomy
  Arms: TLH_plus_PBS
Procedure: TLH _adnexal preservation — TLH without PBS
  Other Names: Standard TLH without salpingectomy
  Arms: TLH _adnexal preservation

SUMMARY:
The aim of this RCT of study is to compare the standard TLH with adnexal preservation with TLH plus prophylactic bilateral salpingectomy (PBS) in terms of ovarian reserve and surgical outcomes

DETAILED DESCRIPTION:
Ovarian cancer accounts for 3% of all female cancers and represents the fifth leading cause of cancer death in the Western world (1). In 90% of cases, these are epithelial ovarian cancers (2).

Because of the biological aggressiveness of this tumor and nonspecific symptoms, that causes a diagnosis at an advanced stage in 75% of cases, ovarian cancer is the gynecological cancer with the highest mortality rate (3).

To date, an effective screening strategy to the early diagnosis of ovarian cancer doesn't exist, so the prophylactic adnexectomy is the only available tool to reduce the incidence and the mortality rate, even if the role of this surgical strategy is controversial, especially in premenopausal women (4). In fact, the American College of Obstetricians and Gynaecologists (ACOG) guidelines recommend the ovarian preservation in premenopausal women with no family history or other risk factors for ovarian cancer (5).

Some clinical studies have shown that the prophylactic adnexectomy and the consequent surgical menopause increase significantly the long term risk of cardiovascular and psychosexual diseases. (6-8). In particular, a case-control study done in a population of 29,380 women subjected to hysterectomy with and without adnexectomy, showed an increased risk of total mortality ( HRs 1.12 95 % CI 1:03 to 1:21 ), lethal and non- lethal cardiovascular disease ( HRs 1.17 95 % CI 1:02 to 1:35 ) and stroke ( HRs 1.14 95 % CI 0.98-1.33 ) (9) . In this population of women subjected to salpingectomy, the surgery wasn't able to lead to an improvement in general survival (10).

Considering the new histopathological classification of the epithelial ovarian cancer, proposed by Kurman (11) and based on new acquisitions about the pathogenesis and the origin of these tumors, it is possible to conceive a new preventive strategy associated with a less morbidity.

In fact, the carcinogenesis model proposed by Kurman, provides for the classification of the most important histological types of epithelial tumors into two types, diversified according to clinico-pathological and genetic features.

The type I is composed of low-grade serous, low-grade endometrioid, clear cell and mucinous carcinomas, whose the ovarian borderline tumors and endometriosis represent the pre-neoplastic lesions. Conversely, the II type includes high-grade endometrioid carcinomas, carcinosarcomas and undifferentiated carcinomas and, more frequently, high-grade serous carcinomas, whose preneoplastic lesion, now, seems to be represented by the serous tubal intraepithelial carcinoma (STIC).

Plenty of evidence, to support the correlation between the epithelial ovarian cancer and the STIC, has been obtained by immunohistochemical and molecular genetics investigations (11). However, from a clinical point of view, this association has been demonstrated only by a study on 55 patients affected by a high-grade serous carcinoma, whose results have shown an involvement in the endosalpinx in 70% of cases and the presence of STIC in about 50% of cases (12).

Some studies, performed on BRCA1 / 2 populations, showed the presence of strongly sites reactive to p53, defined "p53 signature", in the distal tube (13). These sites seem to be more frequent and characteristically multifocal in those tubes with concomitant STIC (14). The finding of "p53 signature" may, therefore, identify an early clonal expansion of the neoplastic proliferation.

This new theory has given the opportunity to prevent this devastating type of cancer by the addition of the prophylactic bilateral salpingectomy (PBS, with the only removal of the tube and the preservation of the ovaries) in all surgical procedures performed in those women with benign diseases once they have accomplished their reproductive desire. The PBS, in place of the current standard procedure (bilateral salpingo-oophorectomy) could reduce the risk of cancer, improving at the same time the quality of life and reducing the risk of premature death due to cardiovascular disease, seen in women subjected to salpingo-oophorectomy before the onset of natural menopause.

Our preliminary data (17) show that, if the bilateral salpingectomy is performed with great care, no patient has negative effects in terms of ovarian function. In addition, in our experience, no perioperative complication is attributable to salpingectomy alone. Despite the retrospective design of our first study, according to the post hoc analysis, these data have shown a significant statistical reliability.

However, prospective data on the effetc of PBS in patients submitted to TLH are still needed

ELIGIBILITY:
Inclusion Criteria:

* Indication to laparoscopic hysterectomy
* Accomplished reproductive desire

Exclusion Criteria:

* Patients with a family history of ovarian cancer and with a known mutation of the BRCA1/2 genes
* Patients with a current or a past history of cancer
* Patients who don't consent to the prophylactic salpingectomy
* Previous adnexal surgery
* PCOS
* Estrogen-progestin therapy in the 2 months prior to the enrollment
* Acute or chronic pelvic inflammatory disorders
* Malignant gynecological neoplasms
* Prior chemotherapy or radiotherapy
* Autoimmune diseases, chronic, metabolic, endocrine and systemic disorders, including hyperandrogenism, hyperprolactinemia, diabetes mellitus and thyroid disease
* Hypogonadotropic hypogonadism
* Taking medications that can cause menstrual irregularities
* Other clinical conditions

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 167 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Ovarian reserve modification | Three months after laparoscopy
  Ovarian reserve modification will be defined as the difference (expressed as Δ) between post-operative and pre-operative values of AMH, FSH, AFC, OV, VI, FI and VFI

SECONDARY OUTCOMES:
Operative time | The same day of surgery
  Time from skin incision to skin closure
variation of hemoglobin level | two hours after the end of surgery
postoperative hospital stay | The day of patient discharge
postoperative return to normal activity | two months after surgery
complication rate | The day of patient discharge

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, Study Director — Magna Graecia University of Catanzaro; Roberta Venturella, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Chair of Obstetrics and Gynecology - University division - UMG, Catanzaro, CZ, Italy

REFERENCES:
- [Background] Morelli M, Venturella R, Mocciaro R, Di Cello A, Rania E, Lico D, D'Alessandro P, Zullo F. Prophylactic salpingectomy in premenopausal low-risk women for ovarian cancer: primum non nocere. Gynecol Oncol. 2013 Jun;129(3):448-51. doi: 10.1016/j.ygyno.2013.03.023. Epub 2013 Apr 2. PMID 23558052